CLINICAL TRIAL: NCT02967445
Title: Physical Examination-Indicated Pessary
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: never started
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2156/15
Record Dates: First submitted 2016-11-11; First posted 2016-11-18 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: PreTerm Birth
MeSH Terms: conditions — Premature Birth | interventions — Cerclage, Cervical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical pessary (Experimental): Arabin Pessary
  Interventions: Device: Arabin Pessary
- Cervical cerclage (Active Comparator): McDonald Cerclage
  Interventions: Device: Cervical cerclage

INTERVENTIONS:
Device: Arabin Pessary — Arabin silicon pessary
  Arms: Cervical pessary
Device: Cervical cerclage
  Arms: Cervical cerclage

SUMMARY:
Cervical insufficiency, previously referred to as cervical incompetence, has classically been defined as painless dilation of the cervix in the absence of contractions or bleeding in the second trimester resulting in recurrent pregnancy losses. Painless mid-trimester cervical dilation is an uncommon finding in the general population occurring in less than 1% of pregnancies. Cerclage for the prevention pregnancy loss in cases with both prior preterm births and/or second trimester losses, as well as second trimester cervical dilatation in the index pregnancy, was first reported in the 1950's. Cerclage placement in this setting has been variably referred to as "physical exam-indicated cerclage", "rescue cerclage", and "emergency cerclage". To date, the benefits of cerclage for this indication are not entirely clear.

A recent meta-analysis showed that physical exam-indicated cerclage is associated with a reduction in perinatal mortality and prolongation of pregnancy when compared to no such cerclage.

Recently, several RCTs have shown that cervical pessary could decrease the incidence of PTB in several populations.

Thus, the aim of our trial as noninferiority trial is to evaluate the efficacy of pessary compared to cervical cerclage in prevention of PTB in women in the setting of mid-trimester cervical dilation

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* Cervical dilation between 1 to 5 cm and/or visible membranes by pelvic exam or speculum exam between at 16-23 6/7 weeks gestation

Exclusion Criteria:

* Pessary or cerclage already in situ
* active vaginal bleeding
* Placenta previa/accreta
* Multiple gestations
* Amniotic membranes prolapsed beyond external os into the vagina, unable to visualize cervical tissue
* Ruptured amniotic membranes at the time of diagnosis of dilated cervix
* Cervical dilation more than 5 cm
* Labor (progressing cervical dilation) or painful regular uterine contractions

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Neonatal survival | From delivery to 28 days

SECONDARY OUTCOMES:
Preterm birth | time of delivery
  <24, <28, <30 weeks. both spontaneous and indicated
Latency | time of delivery
  Time from randomization to delivery
Birth weight | time of delivery
  in grams
gestational age at delivery | time of delivery
  mean of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Napoli, Italy